CLINICAL TRIAL: NCT06387992
Title: Evaluation of the Agreement Between a Consultation With a Nurse Acquiring Three-dimensional Intraoral Images Made With a 3D Intraoral Camera and the Standard Consultation With a Dental Surgeon, in Institutionalized Elderly Subjects
Acronym: GEROdonto3D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PP24023
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Dental Care for Institutionalized Elderly Persons
Keywords: Dental care; oral health; teledentistry; older adults; nursing home

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-dimensional dental acquisition by a nurse (Experimental): Consultation with a trained nurse who will perform a three-dimensional dental acquisition using a 3D intraoral camera
  Interventions: Other: Three-dimensional dental acquisition

INTERVENTIONS:
Other: Three-dimensional dental acquisition — Consultation with a trained nurse who will perform a three-dimensional dental acquisition using a 3D intraoral camera

SUMMARY:
The primary objective of this study will be to assess the agreement between a dental consultation with a nurse acquiring intraoral images, using a 3D intraoral camera, and a standard consultation with a dental surgeon, in institutionalized elderly subjects Institutionalized subjects planned to have a dental consultation and eligible will be included once written informed consent is signed. Their dental consultation will start with a consultation with a nurse to record 3D intraoral images, then a consultation with a dental surgeon for standard dental care, blinded from the nurse consultation will be performed. Thereafter, 3D images will be analyzed by another dental surgeon blinded from the results of both consultations. Agreement on different outcomes between the analysis of the images acquired by the nurse and the standard dental evaluation by a dental surgeon will be assessed.

Agreement on the results between the interpretation of the 3D images acquired by a nurse and the standard consultation by a dental surgeon could lead, in the long term, to a significant step forward in dental care of institutionalized patients.

Indeed, training nursing home nurses to acquire 3D dental images would enable the identification of patients in need of immediate dental care and thus extend the possibilities of access to consultations with a dentist for these patients. This would increase the efficiency of care.

DETAILED DESCRIPTION:
Participation in the study will be offered to any eligible patient in his nursing home prior to his dental consultation. If the patient agrees to participate in the research, he will be included in the study after signing informed consent.

For the included patients, one dental consultation will be planned and organized within the Oral Medicine Unit of the Reims University Hospital. The consultation will be divided into 3 different parts (2 consultations + images analysis):

* 1st part: a consultation with a trained nurse who will perform a three-dimensional dental acquisition using a 3D intraoral camera and who will help the patient complete the General Oral Health Assessment Index (GOHAI)
* 2nd part: a consultation with a dental surgeon, different from the one who analyzes the images. He will perform a standard dental consultation, blinded to the results of the nurse dental consultation.
* 3rd part (without the patient): the three-dimensional images will be interpreted by a dental surgeon (the same for all patients included) blinded to the results of the consultations, in order to obtain the evaluation of the different outcomes. This last step will not require the presence of the patient and can be carried out later.

Participation in the study will not change the patient's dental care.

ELIGIBILITY:
Inclusion criteria:

* Patients institutionalized in one of the nursing homes of the Champagne University Hospital Group in Reims
* Patients who are able to understand and answer questions
* Patients with a planned consultation in the Oral Medicine department of the Reims University Hospital
* Patients affiliated to social security
* Fluent in French
* Patients agreeing to participate in the study

Exclusion criteria:

* Patients who are unable to understand and answer questions
* Totally edentulous patients
* Patients not transportable according to the geriatrician's assessment
* Persons deprived of their liberty by a judicial or administrative decision
* Patients already followed at the Oral Medicine department of the Reims University Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
DMFT index | Day 1
  During dental consultation with a dental surgeon and during the analysis of the 3D images DMFT index (Klein and Palmer, 1940). The index will be assessed from the 3D intraoral images acquired during the nurse consultation and from the standard dental consultation performed by a dental surgeon.
  The DMFT index describes, excluding third molars, the number of teeth:
  * D : Decayed
  * M : missing
  * FT : Filled Teeth The score represents the sum of missing, decayed and/or filled teeth in the same individual. Third molars are not taken into account in the calculation of this score.

SECONDARY OUTCOMES:
Plaque control record | Day 1
  During dental consultation with a dental surgeon and during the analysis of the 3D images Plaque control record (O'Leary et al., 1973). The index will be assessed from the 3D intraoral images acquired during the nurse consultation and from the standard dental consultation performed by a dental surgeon.
  This index records the presence of supragingival plaque on all four tooth surfaces. The result is expressed as a percentage of the number of surfaces with plaque on the total number of faces
General Oral Health Assessment Index (GOHAI) | Day 1
  During the consultation with the nurse The GOHAI assesses self-perceived oral health in older people. It is composed of 12 questions about pain and discomfort, dysfunctions and psychosocial impacts of dental problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France